CLINICAL TRIAL: NCT00116337
Title: Spinal Cord Stimulation to Restore Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Anthony F. Dimarco, Professor of Medicine, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB98-00091; IRB 98-00091; 278855 (Other Grant/Funding Number: Neilsen Foundation)
Record Dates: First submitted 2005-06-28; First posted 2005-06-29 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases; Paralysis; Central Nervous System Diseases; Cough; Trauma, Nervous System; Wounds and Injuries
Keywords: spinal cord injury; paralysis; cough; cervical spinal cord injury; thoracic spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases; Paralysis; Central Nervous System Diseases; Cough; Trauma, Nervous System; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Expiratory Muscle Stimulator (Experimental): Procedure/Surgery: spinal cord stimulation to restore cough
  Interventions: Procedure: Spinal Cord Stimulation to restore cough; Device: Expiratory Muscle Stimulator

INTERVENTIONS:
Procedure: Spinal Cord Stimulation to restore cough — Participants will have small electrodes (metal discs) placed - by a routine surgical procedure - over the surface of their spinal cords on the lower back to stimulate the expiratory muscles and restore cough. These electrodes are then activated at subsequent study visits using the external control unit.
Device: Expiratory Muscle Stimulator — The expiratory muscle stimulator consists of three small electrodes (metal discs) implanted over the surface of their spinal cords on the lower back to stimulate the expiratory muscles and restore cough. These electrodes are connected to an implanted receiver in the abdomen or chest wall. The device is activated through an external antenna connected to an external control box.

SUMMARY:
The purpose of this trial is to determine the efficacy of spinal cord stimulation to produce an effective cough in patients with spinal cord injuries.

DETAILED DESCRIPTION:
Patients with cervical and thoracic spinal cord injuries often have paralysis of a major portion of their expiratory muscles - the muscles responsible for coughing - and therefore, lack a normal cough mechanism. Consequently, most of these patients suffer from a markedly reduced ability to clear airway secretions, a factor which contributes to the development of recurrent respiratory tract infections such as pneumonia and bronchitis. Expiratory muscles can be activated by electrical stimulation of the spinal roots to produce a functionally effective cough.

The purpose of this trial is to determine if electrical stimulation of the expiratory muscles is capable of producing an effective cough on demand. According to the trial researchers, if successful, this technique will prevent the need for frequent patient suctioning - which often requires the constant presence of trained personnel. It will also allow spinal cord injured patients to clear their secretions more readily, thereby reducing the incidence of respiratory complications and associated illness and death.

In the trial, researchers will study 18 adults (18-70 years old) with spinal injuries (T5 level or higher), at least 12 months following the date of injury. After an evaluation of medical history, a brief physical examination, and initial testing, participants will have small electrodes (metal discs) placed - by a routine surgical procedure - over the surface of their spinal cords on the lower back to stimulate the expiratory muscles and restore cough.

ELIGIBILITY:
Inclusion Criteria:

* Stable spinal cord injury T5 level or higher
* Expiratory muscle weakness

Exclusion Criteria:

* Significant cardiovascular disease
* Active lung disease
* Brain disease
* Scoliosis, chest wall deformity, or marked obesity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-09-30 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F. DiMarco, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] DiMarco AF, Romaniuk JR, Supinski GS. Electrical activation of the expiratory muscles to restore cough. Am J Respir Crit Care Med. 1995 May;151(5):1466-71. doi: 10.1164/ajrccm.151.5.7735601.
- [Background] DiMarco AF, Romaniuk JR, Kowalski KE, Supinski G. Pattern of expiratory muscle activation during lower thoracic spinal cord stimulation. J Appl Physiol (1985). 1999 Jun;86(6):1881-9. doi: 10.1152/jappl.1999.86.6.1881. PMID 10368352
- [Background] DiMarco AF, Romaniuk JR, Kowalski KE, Supinski G. Mechanical contribution of expiratory muscles to pressure generation during spinal cord stimulation. J Appl Physiol (1985). 1999 Oct;87(4):1433-9. doi: 10.1152/jappl.1999.87.4.1433. PMID 10517775
- [Background] DiMarco AF, Kowalski KE, Supinski G, Romaniuk JR. Mechanism of expiratory muscle activation during lower thoracic spinal cord stimulation. J Appl Physiol (1985). 2002 Jun;92(6):2341-6. doi: 10.1152/japplphysiol.01231.2001. PMID 12015345
- [Background] Romaniuk JR, Dick TE, Kowalski KE, Dimarco AF. Effects of pulse lung inflation on chest wall expiratory motor activity. J Appl Physiol (1985). 2007 Jan;102(1):485-91. doi: 10.1152/japplphysiol.00130.2006. Epub 2006 Sep 7. PMID 16959914
- [Background] Kowalski KE, Romaniuk JR, DiMarco AF. Changes in expiratory muscle function following spinal cord section. J Appl Physiol (1985). 2007 Apr;102(4):1422-8. doi: 10.1152/japplphysiol.00870.2006. Epub 2006 Dec 7. PMID 17158247
- [Background] DiMarco AF, Kowalski KE, Romaniuk JR. Effects of diaphragm activation on airway pressure generation during lower thoracic spinal cord stimulation. Respir Physiol Neurobiol. 2007 Oct 15;159(1):102-7. doi: 10.1016/j.resp.2007.06.007. Epub 2007 Jun 22. PMID 17681870
- [Background] DiMarco AF, Kowalski KE. Effects of chronic electrical stimulation on paralyzed expiratory muscles. J Appl Physiol (1985). 2008 Jun;104(6):1634-40. doi: 10.1152/japplphysiol.01321.2007. Epub 2008 Apr 10. PMID 18403449
- [Result] DiMarco AF, Kowalski KE, Geertman RT, Hromyak DR. Spinal cord stimulation: a new method to produce an effective cough in patients with spinal cord injury. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1386-9. doi: 10.1164/rccm.200601-097CR. Epub 2006 Mar 16. PMID 16543552
- [Result] DiMarco AF, Kowalski KE, Geertman RT, Hromyak DR, Frost FS, Creasey GH, Nemunaitis GA. Lower thoracic spinal cord stimulation to restore cough in patients with spinal cord injury: results of a National Institutes of Health-Sponsored clinical trial. Part II: clinical outcomes. Arch Phys Med Rehabil. 2009 May;90(5):726-32. doi: 10.1016/j.apmr.2008.11.014. PMID 19406290
- [Result] DiMarco AF, Kowalski KE, Geertman RT, Hromyak DR. Lower thoracic spinal cord stimulation to restore cough in patients with spinal cord injury: results of a National Institutes of Health-sponsored clinical trial. Part I: methodology and effectiveness of expiratory muscle activation. Arch Phys Med Rehabil. 2009 May;90(5):717-25. doi: 10.1016/j.apmr.2008.11.013. PMID 19406289
- [Result] DiMarco AF, Kowalski KE, Hromyak DR, Geertman RT. Long-term follow-up of spinal cord stimulation to restore cough in subjects with spinal cord injury. J Spinal Cord Med. 2014 Jul;37(4):380-8. doi: 10.1179/2045772313Y.0000000152. Epub 2013 Nov 26. PMID 24090524
- [Derived] DiMarco AF, Geertman RT, Nemunaitis GA, Kowalski KE. Impact of the cough stimulation system on the care burden and life quality of caregivers of tetraplegics. J Spinal Cord Med. 2023 Sep;46(5):778-788. doi: 10.1080/10790268.2022.2148845. Epub 2023 Apr 5. PMID 37017634
- [Derived] DiMarco AF, Geertman RT, Nemunaitis GA, Kowalski KE. Comparison of disc and wire electrodes to restore cough via lower thoracic spinal cord stimulation. J Spinal Cord Med. 2022 May;45(3):354-363. doi: 10.1080/10790268.2021.1936388. Epub 2021 Jul 7. PMID 34232841

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were well informed of the details of the study, with particular interest to risks/benefits, and asked to review the Informed Consent before signing.They were given an opportunity to ask questions. Consent was obtained only after all questions and concerns have been addressed.
Groups:
- Clinical Trial - Spinal Cord Stimulation to Restore Cough: Design: Clinical trial. Participants: Subjects with cervical spinal cord injury and weak cough. Interventions: A fully implantable electrical stimulation system was surgically placed in each subject.
Period: Overall Study
Arm/Group | Clinical Trial - Spinal Cord Stimulation to Restore Cough
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Clinical Trial - Spinal Cord Stimulation Cough System: Design: Clinical trial.
  Participants: Subjects with cervical spinal cord injury and weak cough.
  Interventions: A fully implantable electrical stimulation system was surgically placed in each subject.
Arm/Group | Clinical Trial - Spinal Cord Stimulation Cough System
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Overview of study participants
  Participants
    Female | 3
    Male | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 15
  Black or African American | 2

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Expiratory Muscle Activation to Generate Large Airway Pressures Characteristic of Normal Cough.
Description: Airway pressure generation achieved with SCS cough system at the baseline (pre-implant) and 1 year follow up (post-implant).
Time Frame: baseline (pre-implant) and 1 year follow up (post-implant)
Population: Male - 14; Female - 3
Measure: Mean (Standard Error); unit: cmH2O
Groups:
- Pre-Implant - Spontaneous Effort: Airway pressure generation during spontaneous efforts.
- Post-Implantation - Spinal Cord Stimulation (SCS): Changes in airway pressure generation during SCS at the 1-year follow-up.
Arm/Group | Pre-Implant - Spontaneous Effort | Post-Implantation - Spinal Cord Stimulation (SCS)
Number analyzed (Participants) | 17 | 17
cmH2O | 25 (3) | 121 (14)
Statistical Analysis 1: Comparison: Pre-Implant - Spontaneous Effort; Each patient was served as their own control; comparisons was made at various points in the study. Clinical parameters was assessed before the study and also at several end points following the Reconditioning Phase; Test type: Other — Statistical analyses was performed using a repeated measures analysis of variance and Paired t test. A p value of < 0.05 was taken as indicating statistical significance; p < 0.05, ANOVA; Statistical analyses will be performed using a repeated measures analysis of variance and Paired t test

2. Primary Outcome: Effectiveness of Expiratory Muscle Activation to Generate High Peak Airflows Characteristic of Normal Cough.
Description: Peak airflow achieved with SCS cough system at the baseline (pre-implant) and 1 year follow up (post-implant).
Time Frame: baseline (pre-implant) and 1 year follow up (post-implant)
Population: Male - 14; Female - 3
Measure: Mean (Standard Error); unit: L/s
Groups:
- Pre-Implant - Spontaneous Effort: Peak expiratory airflow (L/s) during spontaneous efforts.
- Post-Implantation - Spinal Cord Stimulation (SCS): Changes in peak airflow during SCS at the 1-year follow-up.
Arm/Group | Pre-Implant - Spontaneous Effort | Post-Implantation - Spinal Cord Stimulation (SCS)
Number analyzed (Participants) | 17 | 17
L/s | 1.9 (0.2) | 7.7 (0.9)

3. Secondary Outcome: Incident of Acute Respiratory Tract Infections
Description: The incidence of acute respiratory tract infections, defined by a change in the character, color, or amount of respiratory secretions and requiring antibiotic administration was tracked over the 2-year period prior to implantation of the cough system. The occurrence of respiratory tract infections was determined by subject history and corroborated by review of medical records, when available. After implantation of the cough system, the incidence of acute respiratory tract infections was tracked continually.
Time Frame: baseline (pre-implant) and 1 year follow up (post-implant)
Population: Male - 14; Female - 3
Measure: Mean (Standard Error); unit: Intections per year
Groups:
- Respiratory Tract Infections - Pre-Implant: The incidence of acute respiratory tract infections, defined by a change in the character, color, or amount of respiratory secretions and requiring antibiotic administration was tracked over the 2-year period prior to implantation of the cough system. The occurrence of respiratory tract infections was determined by subject history and corroborated by review of medical records, when available.
- Respiratory Tract Infections - Post-Implant: After implantation of the cough system, the incidence of acute respiratory tract infections was tracked continually.
Arm/Group | Respiratory Tract Infections - Pre-Implant | Respiratory Tract Infections - Post-Implant
Number analyzed (Participants) | 17 | 17
Intections per year | 1.31 (0.32) | 0.29 (0.11)
Statistical Analysis 1: Comparison: Respiratory Tract Infections - Pre-Implant vs Respiratory Tract Infections - Post-Implant; The data prior to implantation were compared with data obtained after implantation of the cough system using a nonparametric analog (Freidman Test) to the standard repeated measures analysis of variance. Statistical significance was assumed at P<0.05. This alpha level was chosen as a correlation for inflated type I error rates because of multiple comparisons. Results are reported as means ± SEs; Test type: Other; p < 0.05, nonparametric analog (Freidman Test)

4. Secondary Outcome: Trained Caregiver Support for Secretion Clearance
Description: The degree of caregiver support was determined as the number of times it was necessary for a caregiver to provide the subject with any form of assistive means of secretion clearance including suctioning, manually assisted cough or use of the insufflation-exsufflation device. Caregiver support was evaluated over a 2-week period prior to implantation of the cough stimulation system and continuously over the course of the initial year and again at the 1-year follow-up.
Time Frame: baseline (pre-implant) and 1 year follow up (post-implant)
Population: Male - 14; Female - 3
Measure: Mean (Standard Error); unit: times/week
Groups:
- Pre-Implant: The degree of caregiver support was determined by the number of times it was necessary for a caregiver to provide the subject with an assistive means of secretion clearance, such as suctioning, manually assisted cough, or insufflation-exsufflation device use. This was determined prospectively over the 2-week period prior to implantation of the cough system
- Post-Implantation - Spinal Cord Stimulation (SCS): The degree of caregiver support was determined by the number of times it was necessary for a caregiver to provide the subject with an assistive means of secretion clearance, such as suctioning, manually assisted cough, or insufflation-exsufflation device use. This was re-evaluated over a 2-week period after implantation of the cough system at the 1-year time points.
Arm/Group | Pre-Implant | Post-Implantation - Spinal Cord Stimulation (SCS)
Number analyzed (Participants) | 17 | 17
times/week | 23.4 (7.3) | 7.7 (4.1)

ADVERSE EVENTS:
Time Frame: 5 year follow up (post-implant)
Groups:
- Post-Implantation - Spinal Cord Stimulation (SCS): Hemodynamic effects: Increases in blood pressure in association with the initial application of SCS.
Arm/Group | Post-Implantation - Spinal Cord Stimulation (SCS)
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-Implantation - Spinal Cord Stimulation (SCS) (N=17)
Infection (Infections and infestations) | 1 (1) — There were no postoperative infections.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-Implantation - Spinal Cord Stimulation (SCS) (N=17)
Hemodynamic effects: Decreases in pulse rate (Nervous system disorders) | 3 (3) — Hemodynamic effects: Decreases in pulse rate in association with the initial application of SCS. With the application of chronic daily stimulation, these changes gradually diminished.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2011-06-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT00116337/Prot_000.pdf
  • Statistical Analysis Plan (2011-06-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT00116337/SAP_001.pdf
  • Informed Consent Form (2011-06-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT00116337/ICF_002.pdf